CLINICAL TRIAL: NCT05191862
Title: An Open-Label, Randomized, Two-Treatment, Two-Sequence, Four-Period, Fully Replicated Crossover Bioequivalence Study of Once Daily PMR Compared to Twice Daily Cilostazol IR Tablets in Healthy Volunteers
Brief Title: Bioequivalence Study of PMR Compared to Cilostazol IR Tablets in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Randomization Error
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GBL21-003
Record Dates: First submitted 2021-12-10; First posted 2022-01-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-04

CONDITIONS: Intermittent Claudication
Keywords: Peripheral Artery Disease; Cilostazol; PMR; Extended-Release Tablet of Cilostazol
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Other): Treatment RTRT
  Interventions: Drug: Cilostazol 100 mg; Drug: PMR 135 mg
- Sequence 2 (Other): Treatment TRTR
  Interventions: Drug: Cilostazol 100 mg; Drug: PMR 135 mg

INTERVENTIONS:
Drug: Cilostazol 100 mg — One Cilostazol 100 mg at 08:00 and another at 20:00, two oral doses (total daily dose of 200 mg)
  Other Names: Treatment R
Drug: PMR 135 mg — Two PMR 135 mg at 08:00, single oral dose (total daily dose of 270 mg)
  Other Names: Treatment T

SUMMARY:
The study is designed to evaluate the bioequivalence and the within-subject variability between the test formulation of extended-release tablet of cilostazol (PMR) administered once daily and the reference formulation of immediate-release tablet of cilostazol (Cilostazol) administered twice-daily in normal healthy male and female subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 to 45 years of age, inclusive, at screening.
* Absence of diseases that could affect the study outcomes.
* Having a body mass index (BMI) between 18.5 and 27.0, inclusive, at screening.
* Females must have a negative serum pregnancy test at screening.
* Understanding and willing to participate in the clinical study and able to comply with study procedures and visits.

Exclusion Criteria:

* History of bleeding tendency.
* Use of anticoagulant agent(s) within one (1) month prior to screening.
* Use of tobacco or nicotine products within six (6) months of screening.
* Intake of over the counter (OTC) or prescription drugs (other than hormonal contraceptives) within two (2) weeks prior to randomization.
* On any investigational drug(s) or therapeutic device(s) within thirty (30) days preceding screening; or anticipating use of any of these therapies during the course of the study (other than the study products).
* History of substance abuse, such as alcohol, IV drugs, and inhaled drugs, within one (1) year prior to screening.
* Known history of having Acquired Immunodeficiency Syndrome (AIDS) or positive pre-study result of infection with Human Immunodeficiency Virus (HIV); known history or positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within three (3) months of screening.
* Positive test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) at any time during the study, either asymptomatic or present with symptoms of Coronavirus disease 2019 (COVID-19).
* Pregnant or breast feeding.
* Women of child-bearing potential not using an effective birth control method. Women of child-bearing potential are defined as women physiologically capable of becoming pregnant, UNLESS they meet the following criteria:

  1. Post-menopausal: 12 months of natural (spontaneous) amenorrhea or less than twelve (12) months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40IU/L, OR;
  2. Six (6) weeks post-surgical bilateral oophorectomy with or without hysterectomy, OR;
  3. Are using one or more of the following acceptable methods of contraception: surgical sterilization (e.g. bilateral tubal ligation, hysterectomy), hormonal contraception (e.g. implantable, injectable, vaginal, patch, and oral), and double-barrier methods. Reliable contraception should be maintained throughout the study and for seven (7) days after study discontinuation.
* Known or suspected hypersensitivity to any ingredient of the study drug(s).
* Donated blood or lost more than 150 mL of blood within three (3) months prior to randomization or plans to donate blood or plasma within four (4) weeks after completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-23 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve, from time zero to last measureable time point (AUC 0-t ) | 0-72 hours after morning dose
AUC from time zero to infinity (AUC 0-∞) | 0-72 hours after morning dose

CONTACTS AND LOCATIONS:
Locations (1):
- Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No